CLINICAL TRIAL: NCT05459389
Title: Efficacy of Early Targeted Antibiotic Therapy in Patients With Sepsis and Septic Shock
Brief Title: Early Targeted Antibiotic Therapy in Patients With Sepsis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rehab Werida (Other)
Responsible Party: Sponsor-Investigator, Rehab Werida, Associate Professor, Damanhour University
Organization: Damanhour University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Early Antibiotic in Sepsis
Record Dates: First submitted 2022-07-12; First posted 2022-07-15 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — Genotype

STUDY DESIGN:
Intervention Model Description: Patients will be randomly allocated to antibiotic regimen guided by conventional culture technique (n=24) or targeted antibiotics therapy guided by resistance genotyping (n=24)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (No Intervention): antibiotic regimen guided by conventional culture technique (n=24)
- Group B (Experimental): targeted antibiotics therapy guided by resistance genotyping (n=24)
  Interventions: Other: targeted antibiotics therapy

INTERVENTIONS:
Other: targeted antibiotics therapy — targeted antibiotics therapy guided by resistance genotyping (n=24)
  Other Names: genotyping
  Arms: Group B

SUMMARY:
The aim of this study is to assess the efficacy of early targeted antibiotic therapy in patients with sepsis and septic shock using the new biomarker Sirtuin 1 and PCR for bacterial resistance detection.

The primary outcome is change in SOFA score (ΔSOFA) which will be calculated by subtracting the final SOFA score and sirtuin 1 level at 5 days from the corresponding initial value at enrollment.

Secondary outcomes included mortality rates, ventilator free days and length of icu stay.

DETAILED DESCRIPTION:
* A prospective, single-center, open labeled, randomized interventional study
* Patients will be recruited from a private hospital in Alexandria
* Approval will be obtained from Research Ethics Committee of Faculty of Pharmacy, Damanhour University
* Fourty eight critically ill patients, with sepsis and septic shock according to the 2016 third international consensus definitions, will be included
* Patients with risk for Carbapenemase producing organisms:

  * Use of broad spectrum cephalosporins and/or carbapenems within the past three months
  * Polytrauma
  * Diabetes
  * Malignancy
  * Organ transplantation
  * Mechanical ventilation
  * Indwelling urinary or venous catheters
  * Overall poor functional status or severe illness
  * Residence in a long-term care facility(18-28).
* The baseline characteristics of the patients will be collected at the time of enrollment. The collected data included age, sex, ratio of septic shock to sepsis, ratio of ventilated to non-ventilated patients, source of infection, vital signs, laboratory data, arterial blood gas (ABG), APACHE II score, Glasgow Coma Scale score, and SOFA scores. The level of Procalcitonin (PCT) and Sirtuin-1 will also be measured at this time(29).
* Patients will be randomly allocated to antibiotic regimen guided by conventional culture technique (n=24) or targeted antibiotics therapy guided by resistance genotyping (n=24) (29, 30).
* Levels of Sirtuin1 will be detected using ELISA kits as prescribed by manufacturer.
* Traditional diagnostic microbiology techniques relying on the growth of organisms on appropriate culture media (Control group).
* Qualitative Multiplex pcr test will be used for rapid detection of carbapenemases genes (Intervention group)
* Statistical tests appropriate to the study will be conducted to evaluate significance of results
* Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years or older
2. A definite diagnosis of sepsis or septic shock according to the definition of the 2016 SCCM/ESICM task force.
3. Patients at risk for carbapenemase producing organisms

Exclusion Criteria:

1. Pregnant and lactating women
2. hematological disorders (e.g., leukemia, myelodysplastic syndrome, neoplastic metastases to bone marrow),
3. life-threatening diseases (e.g., malignant solid tumors), acquired immunodeficiency syndrome.
4. Lethal traumatic injury
5. Acute Physiologic Assessment and Chronic Health Evaluation II (APACHE II) score ≥34 (due to high predicted mortality of 80%)
6. Primary fungal or viral infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Sirtuin1 (ng/ml) | 5 days
  Levels of Sirtuin1 will be detected using ELISA kits as prescribed by manufacturer.
SOFA (score) | 5 days
  SOFA score (ΔSOFA) which will be calculated by subtracting the final SOFA score at 5 days from the corresponding initial value at enrollment.

SECONDARY OUTCOMES:
mortality rates (%) | 5 days
  number of dead patients.
ventilator free days (days) | 5 days
  count of days free from ventilator,
length of icu stay (Days) | 5 days
  count of days in ICU

CONTACTS AND LOCATIONS:
Overall Officials: Rehab H Werida, Ass. Prof., Study Director — Damanhour University; Noha Elbassiony, Principal Investigator — Damanhour University; Eman Momtaz, Principal Investigator — Damanhour University
Locations (1):
- Rehab Hussein Werida, Damanhūr, Elbehairah, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singer M, Deutschman CS, Seymour CW, Shankar-Hari M, Annane D, Bauer M, Bellomo R, Bernard GR, Chiche JD, Coopersmith CM, Hotchkiss RS, Levy MM, Marshall JC, Martin GS, Opal SM, Rubenfeld GD, van der Poll T, Vincent JL, Angus DC. The Third International Consensus Definitions for Sepsis and Septic Shock (Sepsis-3). JAMA. 2016 Feb 23;315(8):801-10. doi: 10.1001/jama.2016.0287. PMID 26903338
- [Result] Martinez ML, Plata-Menchaca EP, Ruiz-Rodriguez JC, Ferrer R. An approach to antibiotic treatment in patients with sepsis. J Thorac Dis. 2020 Mar;12(3):1007-1021. doi: 10.21037/jtd.2020.01.47. PMID 32274170
- [Result] Bhattacharyya RP, Bandyopadhyay N, Ma P, Son SS, Liu J, He LL, Wu L, Khafizov R, Boykin R, Cerqueira GC, Pironti A, Rudy RF, Patel MM, Yang R, Skerry J, Nazarian E, Musser KA, Taylor J, Pierce VM, Earl AM, Cosimi LA, Shoresh N, Beechem J, Livny J, Hung DT. Simultaneous detection of genotype and phenotype enables rapid and accurate antibiotic susceptibility determination. Nat Med. 2019 Dec;25(12):1858-1864. doi: 10.1038/s41591-019-0650-9. Epub 2019 Nov 25. PMID 31768064